CLINICAL TRIAL: NCT01697540
Title: Tropical Medicine Center (TMC), Kaohsiung Medicine University Hospital (KMUH)
Brief Title: Management of Highly Active Anti-retroviral Therapy-related Hyperlipidemia Among HIV-infected Patients in Taiwan
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-2012-05-05(I)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2017-01

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
1. Written informed consent must be obtained before any study specific procedures are undertaken.
2. The process of the experiment (brief describe) The patients must come back for follow during 4 to 12 weeks after starting the new therapy. The investigators will follow the patients' lipid profile and any side effects and stop the observation till 36 months after starting the new therapy. The serum level of HIV-VL, CD4, GOT, GPT, triglyceride, cholesterol, HDL-cholesterol, and LDL-cholesterol will be checked every 3 months. The patients' chart and all data will be delinked to protect the patients' right and privacy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients who receive HAART therapy but have metabolic side effects.
* Age over 20 years old

Exclusion Criteria:

* Abnormal liver function: GOT or GPT 5 times over normal upper limit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV/AIDS group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical medicine center, Kaohsiung City, Taiwan